CLINICAL TRIAL: NCT00084643
Title: A Phase I Study of GTI-2040 in Combination With Oxaliplatin and Capecitabine in Patients With Advanced Metastatic Solid Tumors
Brief Title: GTI-2040, Oxaliplatin, and Capecitabine in Treating Patients With Locally Advanced or Metastatic Colorectal Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03077; PHI-41; U01CA062505 (NIH); CDR0000365466 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — GTI2040; Oxaliplatin; Capecitabine

ARMS (1):
- Treatment (GTI-2040, capecitabine, oxaliplatin) (Experimental): Patients receive GTI-2040 IV continuously on days 1-14, oral capecitabine twice daily on days 2-15, and oxaliplatin IV over 2 hours on day 2 of the first course. In all subsequent courses, capecitabine is administered on days 1-14, oxaliplatin is administered on day 1, and GTI-2040 is administered as in course 1. Courses repeat every 21 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Biological: GTI-2040; Drug: oxaliplatin; Drug: capecitabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: GTI-2040 — Given IV
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of capecitabine when given together with GTI-2040 and oxaliplatin in treating patients with locally advanced or metastatic colorectal cancer or other solid tumors. Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. GTI-2040 may increase the effectiveness of chemotherapy by making tumor cells more sensitive to the drugs. Giving GTI-2040 together with oxaliplatin and capecitabine may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated (MTD) of a 21 day cycle of capecitabine given orally twice daily for 14 days in combination with oxaliplatin given intravenously on day 1 and GTI-2040 given as a continuous infusion over 14 days in patients with advanced metastatic solid tumors.

II. To describe the toxicities at each dose level studied.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of GTI-2040, capecitabine, and oxaliplatin when these are given in combination.

II. To evaluate levels of ribonucleotide reductase -M2 subunit (RR-M2) mRNA levels using TaqMan RT-PCR in peripheral blood mononuclear cells and in tumor samples (when available). TRF support will be required and sought.

III. To quantitate changes in dCTP levels in peripheral blood mononuclear cells during treatment as a surrogate marker of RR inhibition. TRF support will be required and sought.

OUTLINE: This is a multicenter, dose-escalation study of capecitabine.

Patients receive GTI-2040 IV continuously on days 1-14, oral capecitabine twice daily on days 2-15, and oxaliplatin IV over 2 hours on day 2 of the first course. In all subsequent courses, capecitabine is administered on days 1-14, oxaliplatin is administered on day 1, and GTI-2040 is administered as in course 1. Courses repeat every 21 days in the absence of disease progression and unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced or metastatic colorectal cancer that is not amenable to surgical treatment; selected patients with advanced disease in incurable cancers of other types may be considered
* Patients must have histological or cytological proof of malignancy
* Patients must have had at least one standard prior chemotherapy for locally advanced or metastatic disease with no prior oxaliplatin containing regimen; patients who relapse within 12 months of adjuvant therapy are eligible
* Karnofsky performance status of >= 60%
* Absolute neutrophil count > 1500/ul
* Platelets > 100,000/ul
* Total bilirubin within institutional normal limits
* AST (SGOT)/ALT (SGPT) within 2.5 x institutional normal limits
* Alkaline phosphatase within 2.5x institutional normal limits
* Creatinine within institutional normal limits or a calculated creatinine clearance > 60 ml/min
* Patients should have no greater than grade 1 neuropathy (CTCAE v3.0)
* Ability to understand and the willingness to sign a written IRB approved consent document
* Measurable disease not required
* Previous chemotherapy must have been completed > 21 days before treatment on this study (> 6 weeks for mitomycin-c or nitrosoureas)
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Active or chronic hepatitis B or C
* HIV positive patients receiving antiviral therapy because of possible pharmacokinetic interactions
* Uncontrolled intercurrent illnesses including but not limited to ongoing or active infections, symptomatic congestive heart failure, unstable angina, or cardiac arrhythmia
* Pregnant or nursing women are excluded due to the potential for teratogenic effects and for potential deleterious effects on the infant; woman of childbearing age and men must practice an effective form of contraception
* Patients with known brain metastasis are excluded due their poor prognosis and due to possible neurologic sequelae that could confound the evaluation of the investigational treatment
* Patients requiring anticoagulation are excluded as polyanions are known to inhibit clotting mechanisms and phosphorothioate oligonucleotide may act in a similar mechanism; patients receiving low dose prophylactic Coumadin (1 mg/day) may be included
* Medical, social, of psychological factors that would interfere with consent and follow-up
* Patients with a diagnosis of pulmonary fibrosis or a pulmonary interstitial process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
MTD of the combination of GTI-2040, oxaliplatin and capecitabine based on the incidence of dose-limiting toxicity (DLT) as assessed by CTCAE version 3.0 | 21 days
  Adverse events will be summarized by grade, attribution, and organ system. Hematological and clinical chemistry laboratory results will be included in the adverse event summary.

SECONDARY OUTCOMES:
Objective response (confirmed PR and CR) according to RECIST | At 6 weeks
  Calculated with exact binomial 95% confidence interval.
Pharmacokinetics | At baseline, and at 7 and 14 days after the start of infusion
  Peak and integrated blood levels will be summarized by dose level, and displayed in scatterplots with RR-M2 mRNA levels and changes.
Change in biochemical and molecular correlates | From baseline to up to 4 years
  Molecular correlates will be analyzed descriptively in relation to clinical outcome. The association with progression-free survival or overall survival will be assessed by dichotomizing the measures of gene expression at the median (or by previously-established cut-points) and constructing Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shibata, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States